CLINICAL TRIAL: NCT04364048
Title: Induction Durvalumab Followed by Chemoradiation and Consolidation Durvalumab (MEDI4736) for Stage III Non-small Cell Lung Cancer
Brief Title: Durvalumab Followed by Chemoradiation and Consolidation Durvalumab for Stage III Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study enrollment was halted due to pandemic-related slow accrual
Sponsor: Rachel Sanborn (Other)
Collaborators: AstraZeneca (Industry); Providence Cancer Center, Earle A. Chiles Research Institute (Other)
Responsible Party: Sponsor-Investigator, Rachel Sanborn, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN18-357
Record Dates: First submitted 2020-04-24; First posted 2020-04-27 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Non-small Cell Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — durvalumab; Drug Therapy; Cisplatin; Carboplatin; Etoposide; Pemetrexed; taxane; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Induction durvalumab, chemoradiation, consolidation durvalumab (Experimental): Induction durvalumab at 1500 mg intravenously (IV) on Day 1 of a four week cycle for 1 cycle, followed by concurrent definitive chemoradiation, followed by consolidation durvalumab at 1500 mg IV Day 1 of every 4 week cycle for up to 12 cycles.
  Interventions: Drug: Induction Durvalumab; Drug: Chemotherapy; Radiation: Radiation; Drug: Consolidation durvalumab

INTERVENTIONS:
Drug: Induction Durvalumab — Induction durvalumab at 1500 mg intravenously (IV) will be given on Day 1 of a four week cycle for 1 cycle,
  Other Names: IMFINZI
Drug: Chemotherapy — Concurrent chemoradiation will be with platinum-based chemotherapy (cisplatin or carboplatin, with etoposide, taxane, or pemetrexed) selected at the treating physician's discretion. The chemotherapy regimen used should be administered per institutional standards following the prescribing guidelines for each drug
  Other Names: cisplatin; carboplatin; etoposide; pemetrexed; taxane
Radiation: Radiation — Treatment will be delivered using IMRT or 3DCRT using typically 6-10MV photons per institutional standards. 4D simulation and appropriate IGRT are encouraged. Radiation therapy must begin within one week of the first day of chemotherapy (or vice versa). Therapy will be 1.8-2 Gy per day; 5 days per week, excluding holidays per institutional standard as this is a standard of care regimen for this patient population. 54-66 Gy will be delivered.
Drug: Consolidation durvalumab — Durvalumab at 1500 mg intravenously (IV) will be given on Day 1 of a four week cycle for 12 cycles
  Other Names: IMFINZI

SUMMARY:
Single arm study of induction durvalumab (1500 mg IV) for 1 cycle (every 4 weeks), administered prior to starting concurrent definitive chemoradiation, followed by consolidation durvalumab (1500 mg IV every 4 weeks) for up to 12 cycles.

The study will include an initial safety run-in portion. Patients in the safety run-in will be monitored through completion of induction durvalumab, chemoradiation, and 2 cycles of consolidation durvalumab for assessment of safety prior to completion of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0 or 1.
* Histological or cytological confirmation of stage III non-small cell lung cancer per AJCC, 8th edition, eligible for curative-intent concurrent chemoradiation. NOTE: subjects are not candidates for surgical resection either due to medical inoperability or surgically unresectable disease.
* Measurable disease according to RECIST 1.1 criteria.
* Plan for treatment with concurrent chemoradiation with a dose of radiation ranging from 54-66 Gy:

  * Planned mean dose delivery to the lung <20 Gy
  * V20 <35%
* No prior therapy for stage III NSCLC.
* Demonstrate adequate organ function as defined in the protocol. All screening labs to be obtained within 14 days prior to registration.
* Females of childbearing potential must have a negative serum pregnancy test within 24 hours of C1D1. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential must be willing to abstain from heterosexual intercourse or to use contraception as outlined in the protocol.
* Men who are sexually active with WOCBP must be willing to abstain from heterosexual intercourse or to use contraception as outlined in the protocol.
* Life expectancy of at least 12 weeks per investigator discretion.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

* Prior therapy for stage III NSCLC
* Mixed histology with small cell lung cancer will not be allowed.
* Sequential chemoradiation will not be permitted.
* Induction and consolidation chemotherapy (separate from concurrent chemoradiation) will not be allowed.
* Prior exposure to anti-PD-1 or anti-PD-L1 antibodies including durvalumab.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* History of pulmonary fibrosis, interstitial lung disease, or pneumonitis requiring steroids.
* Active or prior documented autoimmune disease within the last 2 years. Patients with vitiligo, stable hypothyroidism, Grave's disease, or psoriasis not requiring systemic treatment are not excluded.
* Body weight < 30 kg
* Active and ongoing steroid use, except for non-systemically absorbed treatments (such as inhaled or topical steroid therapy for asthma, COPD, allergic rhinitis).
* Active infection requiring systemic therapy.
* Uncontrolled current illness that in the opinion of the investigator renders the investigational treatment plan unsafe.
* Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. NOTE: Local surgery of isolated lesions for palliative intent is acceptable.
* Active other malignancy; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Treatment with any investigational drug within 30 days prior to registration.
* History of organ transplantation (including allogeneic stem cell transplantation).
* Other medical or psychiatric conditions that in the opinion of the site investigator would preclude safe participation in this protocol.

Eligibility Criteria for Consolidation Durvalumab

* Patients must have recovered from toxicities associated with prior chemoradiation to CTCAE < Grade 2.
* Patients must not have progressed following chemoradiation therapy, as measured on imaging per RECIST 1.1.
* Confirmation of ECOG Performance Status of 0 or 1.
* Any grade pneumonitis from prior chemoradiation will not be permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Sanborn, MD, Principal Investigator — Providence Cancer Institute
Locations (5):
- United States (5):
  - Rush University Medical Center, Chicago, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - HealthPartners Institute, Minneapolis, Minnesota
  - Summit Medical Group, P. A., Berkeley Heights, New Jersey
  - Providence Portland Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 67 [55 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Histology at Study Entry [Count of Participants; unit: Participants]
  Adenocarcinoma | 4
  Adenosquamous | 1
  Squamous | 5

OUTCOME MEASURES:

1. Primary Outcome: 12-Month Progression Free Survival (PFS)
Description: 12-month progression-free survival will be measured using imaging after completion of chemoradiation, prior to C1 consolidation durvalumab (1-42 days after completion of chemoradiation) per RECIST 1.1.
  RECIST 1.1 Criteria for Response are:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: From the time of treatment initiation until progression, up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab
Number analyzed (Participants) | 10
percentage of participants | 30 [11.6 to 77.33]

2. Primary Outcome: Evaluate the Safety and Feasibility of Induction Durvalumab Using NCI CTCAE v5.0 for Toxicity Grading.
Description: All subjects receiving at least one dose of durvalumab will be evaluable for toxicity. The National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, will be used for toxicity grading. Please refer to the study calendar for the schedule of toxicity assessment.
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab
Number analyzed (Participants) | 10
participants
  Anemia | 2
  Neutropenia | 3
  Thrombocytopenia | 1
  Alkaline Phosphate Increased | 1
  Anorexia | 1
  Anxiety | 1
  Chills | 1
  Constipation | 1
  Creatinine Increase | 1
  Diarrhea | 1
  Dizziness | 1
  Dyspnea | 2
  Fever | 1
  Hiccups | 1
  Hyperkalemia | 1
  Hypomagnesemia | 1
  Hypothyroidism | 1
  Infusion Reaction | 1
  Insomnia | 1
  Mucositis/Mouth Pain | 2
  Odynophagia | 1
  Pruritis | 1
  Rash | 5
  Neuropathy | 1

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR will be measured using two timepoints, per RECIST 1.1. "ORR1" will be assessed using baseline imaging in comparison to imaging obtained after completion of induction durvalumab and chemoradiation. "ORR2" will be assessed using imaging after completion of induction durvalumab and chemoradiation in comparison to imaging obtained while receiving, and after completion of, consolidation durvalumab.
  RECIST 1.1 Criteria for response are as follows:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab
Number analyzed (Participants) | 10
Participants
  Complete Response | 2
  Partial Response | 5
  Stable Disease | 3

ADVERSE EVENTS:
Time Frame: From initiation of subject consent until off study, up to 3.5 years.
Arm/Group | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab
All-Cause Mortality (participants affected / at risk) | 3/10
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab (N=10)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Durvalumab, Chemoradiation, Consolidation Durvalumab (N=10)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Creatinine Increase (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Infusion Reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Mucositis/Mouth Pain (Gastrointestinal disorders) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Neuropathy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT04364048/Prot_SAP_000.pdf